CLINICAL TRIAL: NCT00001531
Title: Potential Role of CMV in Restenosis Following Angioplasty, in Atherosclerosis, and in Endothelial Dysfunction
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 960099; 96-H-0099
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-08

CONDITIONS: Arterial Occlusive Diseases; Atherosclerosis; Coronary Disease; Cytomegalovirus Infections
Keywords: Atherogenesis; Cell Mediated Immunity; Coronary Artery Disease
MeSH Terms: conditions — Arterial Occlusive Diseases; Atherosclerosis; Coronary Disease; Cytomegalovirus Infections; Coronary Artery Disease

SUMMARY:
The purpose of this study is to investigate whether the susceptibility of subjects to atherosclerosis is influenced by prior CMV exposure, whether the susceptability to endothelial dysfunction in patients with and in patients without atherosclerosis is influenced by prior CMV exposure.

DETAILED DESCRIPTION:
The purpose of this study is to investigate whether the susceptibility of subjects to atherosclerosis is influenced by prior CMV exposure, whether the susceptability to endothelial dysfunction in patients with and in patients without atherosclerosis is influenced by prior CMV exposure.

ELIGIBILITY:
Patients who are being evaluated to determine if they have CAD or those who have already been studied and the presence or absence of CAD has been ascertained.

No patients who have not been evaluated for CAD.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 355
Dates: Start 1996-06; Study Completion 2000-09

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Speir E, Modali R, Huang ES, Leon MB, Shawl F, Finkel T, Epstein SE. Potential role of human cytomegalovirus and p53 interaction in coronary restenosis. Science. 1994 Jul 15;265(5170):391-4. doi: 10.1126/science.8023160.
- [Background] Schrier RD, Freeman WR, Wiley CA, McCutchan JA. Immune predispositions for cytomegalovirus retinitis in AIDS. The HNRC Group. J Clin Invest. 1995 Apr;95(4):1741-6. doi: 10.1172/JCI117851. PMID 7706482